CLINICAL TRIAL: NCT00011336
Title: Prospective Cohort Study of Respiratory Function and Illness in Chronic SCI
Brief Title: Determine the Association Between the Level of SCI With Chronic Respiratory Symptoms, Measures of Pulmonary Function, and Respiratory Illness.
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 717B
Record Dates: First submitted 2001-02-15; First posted 2001-02-19 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2003-02

CONDITIONS: Spinal Cord Injuries
Keywords: SCI; chronic respiratory symptoms; measures of pulmonary function; respiratory illness
MeSH Terms: conditions — Spinal Cord Injuries

SUMMARY:
This study is using a standardized method to assess respiratory function in SCI in order to determine the association between level of SCI with chronic respiratory symptoms, measures of pulmonary function, and respiratory illness, both cross-sectionally and longitudinally.

DETAILED DESCRIPTION:
Primary Objectives: Determine the association between level of spinal cord injury (SCI) with chronic respiratory symptoms, measures of pulmonary function, and respiratory illness, both cross-sectionally and longitudinally.

Intervention: None

Study Abstract: This study is using a standardized method to assess respiratory function in SCI in order to determine the association between level of SCI with chronic respiratory symptoms, measures of pulmonary function, and respiratory illness, both cross-sectionally and longitudinally.

A community-based mail survey was made of 1147 subjects (42% response rate; 2 mailings, n=485). Additional subjects injured >1 year ago underwent testing at the West Roxbury VAMC (FVC, FEV1, TLC and subdivisions, maximal inspiratory and expiratory pressures (MIP/MEP), and completed a health questionnaire based on the ATS DL-78 respiratory questionnaire. Between 10/94-9/98, a cross-sectional cohort of 361 subjects with chronic SCI were tested. Multiple logistic regression was used to examine predictors of respiratory symptoms and chest illness determined from the questionnaire.

From the community-based mail survey, SCI with complete cervical injury (CC) the odds reporting ?any wheeze? relative to lower SCI levels (odds ratio (95%CI)) was 3.34 (1.75-6.40), p<0.001, and for ?persistent wheeze? was 2.41 (1.11-5.22), p=0.023. The odds of reporting chronic cough or phlegm were not increased (p=0.40 and 0.07 respectively). Active cigarette smoking was the strongest predictor of respiratory symptoms. In a subset of subjects tested at our VAMC, the odds of CC SCI of reporting chest illness resulting in time off work, indoors at home, or in bed over 3 years before questionnaire completion relative to incomplete injury was 3.00 (1.12-8.01), p=0.029. For 1 PPD current smokers the risk of chest illness was 3.91 (1.71-8.95), p=0.001, for subjects who smoked post injury but quit within the previous 10 years the odds was 3.00 (1.00-8.97), p=0.05. For other former smokers the odds were not significantly increased. Subjects who reported ?persistent wheeze? were nearly 3 times as likely to have reported a chest illness (p=0.036). After using a wheelchair, 31% of CC subjects reported breathlessness, compared to 15% with complete high thoracic, and 11% of lower injuries (p=0.04 trend). Subjects who were not wheelchair athletes, even when lung function and SCI level were noted, were twice as likely not to report breathlessness compared to athletes (p=0.032). Subjects with SCI were able to produce reproducible spirometry. Analysis of the effect of SCI level on lung function is in progress, as are analyses examining predictors of chest illness in the workers tested to date.

We have developed a method to assess respiratory function in SCI. Using these methods, complete cervical SCI have been found to experience more wheeze and breathlessness than others with SCI, and are more likely to report a chest illness. However, active cigarette smoking was the most important predictor of chest illness and respiratory symptoms rather than injury level or completeness. Therefore, it is likely that SCI based smoking cessation programs would result in significantly reducing respiratory morbidity in this population. The introduction of exercise programs might also result in a decreased prevalence of breathlessness in complete cervical SCI.

ELIGIBILITY:
Spinal cord injury of >= 1 year in duration, and no other neuromuscular diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 1998-07; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Overall Officials: Robert Brown, MD, Study Director; Carlos Tur, MD, Study Director
Locations (1):
- Boston VA Health Care System, West Roxbury, Massachusetts, United States